CLINICAL TRIAL: NCT05111964
Title: A Pilot Study in High Intensity Focused Ultrasound Ablation of Soft Tissue Sarcoma and Small Symptomatic Desmoid Tumours
Brief Title: HIFU Ablation of Soft Tissue Sarcoma
Acronym: SarcAblate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Surgical Intervention Trials Unit, Oxford, UK (Unknown); National Institute for Health Research, United Kingdom (Other Government); Oxford Radiology Research Unit, Churchill Hospital, Oxford, UK (Unknown)
Responsible Party: Principal Investigator, Paul Lyon, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15182
Record Dates: First submitted 2021-10-11; First posted 2021-11-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma; Desmoid Tumors
Keywords: HIFU; Focused Ultrasound; Immunology
MeSH Terms: conditions — Sarcoma; Desmoid Tumors | interventions — High-Intensity Focused Ultrasound Ablation

STUDY DESIGN:
Intervention Model Description: No randomisation. Four recruitment cohorts, patients with:
  1. Soft tissue sarcoma 1-5cm for resection
  2. Soft tissue sarcoma >1cm with infield recurrence for resection
  3. Soft tissue sarcoma unsuitable for resection or further chemo- or radiotherapy
  4. Small (1-8 cm) symptomatic desmoid tumour unsuitable for surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIFU Treatment of STS or Intra-abdominal Desmoid Tumour (Experimental): All participants receive HIFU to their target tumour, hence this is a single arm study with 4 recruitment pathways.
  Interventions: Device: High Intensity Focused Ultrasound Ablation; Diagnostic Test: Tumour Biopsy and Venous Blood Tests

INTERVENTIONS:
Device: High Intensity Focused Ultrasound Ablation — The focused ultrasound exposure will be performed using the Haifu® Model-JC200 Focused Ultrasound Tumour Therapeutic System at the Churchill Hospital site, CE-approved for tumour therapy (or subsequent CE-approved device upgrades by Haifu®), the device completely upgraded in 2025. The participant will be positioned over the therapeutic device and water bath used to transmit the focused ultrasound to the target tumour. No anaesthesia or any combination of local anaesthesia, nerve block, epidural, conscious sedation or general anaesthetic may be used, depending on anatomical location, size of tumour, preference of HIFU team, patient and anaesthetist and other patient factors.
  In therapy mode, the tumour volume is treated with focused ultrasound to ablate the tumour tissues to high temperatures (in excess of 60ºC) using focused ultrasound targeted from outside the body.
  Patients are typically discharged with 24 hours.
Diagnostic Test: Tumour Biopsy and Venous Blood Tests — Where appropriate, participants are also encouraged to undergo a pre-HIFU (and in the case of unresectable STS, post-HIFU) ultrasound biopsy of the target tumour and additional blood tests to inform the immunological aspects of the study. Having the biopsy does not mandate enrolment on the trial, and patients will be free to leave the trial at any stage. The pre-HIFU (and post-HIFU) biopsies are altruistically encouraged but not absolutely essential to enrolment on the trial.
  Biopsies will be performed under ultrasound guidance by an experienced radiologist using local anaesthetic.

SUMMARY:
Around 3,300 people are diagnosed with soft tissue sarcoma (STS) each year in the UK, and a significant proportion of STS diagnoses are in people aged under 30 years. STS can arise from various tissue types and is comprised of over 50 tumour types. Although STS is treated with a combination of surgery, radiotherapy and chemotherapy, the prognosis is relatively poor with a five-year survival rate of 54%. There is an unmet need for further treatment modalities in STS.

High intensity focused ultrasound (HIFU) is a non-invasive way of treating cancers with minimal side effects, low complication rate and quick recovery. Ultrasound waves are used to destroy tumour cells and improvements in technology and experience are enabling complete destruction of tumour. HIFU also releases tumour antigens, increasing the immune response against cancer. HIFU has received FDA approvals for several indications, including bone metastases and we are using a CE-approved HIFU device in Oxford (UKCA-approvals anticipated for 2023). There have been some publications from China showing promise in STS, however this technology needs further evaluation within the UK's healthcare setting.

This study will recruit patients with both resectable and unresectable STS, in addition to unresectable small symptomatic desmoid tumours. 12-16 patients, and a minimum of 10 patients with malignant STS, will be treated over a maximum recruitment period of three years. HIFU treatment will be carried out as a day case procedure, and patients will be expected to be discharged home the same day.

The study is designed to generate evidence regarding safety and feasibility of HIFU for ablation of STS and intra-abdominal desmoids. In addition, the study is anticipated to provide information about the efficacy of HIFU against these tumour types which can help in the design of later phase studies. Short-term outcomes include feasibility, safety and the completeness of destruction of the tumour. Long-term outcomes include one-year survival, local recurrence and quality of life metrics (including pain scores). The study will also look at immunological response following ablation of STS using both blood and tumour samples pre- and post-HIFU ablation.

DETAILED DESCRIPTION:
Tissues that can be affected by soft tissue sarcomas include fat, muscle, blood vessels, nerves, deep skin tissues, tendons and ligaments. Sarcoma accounts for 1% of all cancer diagnoses; around 3,300 people are diagnosed with soft tissue sarcoma (STS) each year in the UK. The incidence of STS is unusual for cancer in that a relatively large proportion can occur in children and young adults, with 9% of cases in the under 30-year group and only 43% of cases in the 65 and over group. Whilst STS is rare, it remains a significant cause of morbidity and mortality. Prognosis is typically poor, with a five-year overall survival of approximately 54%.

The Oxford Bone and Soft Tissue Tumour Service at the Nuffield Orthopaedic Centre, Oxford, is a nationally approved tertiary referral centre for the treatment of soft tissue and primary bone sarcomas, receiving 400 new patient referrals annually. These patients are currently treated via a multidisciplinary approach involving expert radiologists, surgeons, clinical oncologists and histopathologists.

At our centre, patients with smaller (<5cm) STS proceed directly to surgical resection; this provides a low-risk opportunity to evaluate safety, feasibility and efficacy of novel pre-operative non-ionising ablative technologies, such as High Intensity Focused Ultrasound (HIFU). Patients with larger (>5cm) resectable STS currently receive neoadjuvant radiotherapy within six weeks of surgery, in line with national guidelines (Dangoor, 2016). Upon recurrence within the radiotherapy field (in-field recurrence), radiotherapy has high morbidity, including complications such as poor wound healing and infection (Tsagozis, 2018), and is not indicated prior to further surgical resection. Thus, in resectable cases of in-field recurrence, there is further opportunity to evaluate non-invasive HIFU, anticipated to both reduce tumour size and tumour vascularity, facilitating subsequent surgical resection. Furthermore, recurrent STS or metastatic STS not suitable for surgery have limited treatment options, and if not suitable for further chemo- or radio-therapy, HIFU may provide an alternative treatment option before palliation.

HIFU is a versatile treatment modality capable of destruction of tumours by focusing ultrasound waves from outside the body, usually through the medium of water, to cause ablation at a precise anatomical location.

It has demonstrated an impressive safety profile by virtue of being both non-invasive and lacking radiation, leading to FDA approvals for several indications including pain relief in bone metastases (Scipione, 2018) and uterine fibroids. Previous studies using an ultrasound-guided therapeutic device in China have demonstrated that HIFU is a successful treatment modality for soft tissue sarcoma (Yu, 2019), but this treatment has currently not been widely investigated within the UK's health care setting.

The University of Oxford and the Oxford University Hospitals NHS Trust have extensive clinical HIFU experience. The first extracorporeal HIFU device in Europe was used for a study performed at the Churchill Hospital between 2002 and 2004 (Illing, 2005). The study used an ultrasound-guided HIFU system (Model-JC Tumour Therapy System, HAIFU Technology Company Ltd, Chongqing, China) to treat 30 patients with tumour deposits in the kidney or liver and demonstrated both safety and efficacy. This was followed by a non-randomised Phase II clinical trial of HIFU ablation of liver tumours (Leslie, 2008), which compared radiological response against histological findings and again demonstrated safety and feasibility for non-invasive treatment of solid tumour deposits. These studies have led to CE-marking of the JC and JC-200 treatment devices for non-invasive treatment of solid tumours such as liver cancer, kidney tumours, breast cancer, bone tumours, pancreatic tumours and uterine fibroids, based on previous clinical trials at our unit (Lyon, 2019), the latter indication recently receiving NICE approval for US-guided HIFU ablation.

Safety and efficacy of HIFU has already been demonstrated for sacral chordoma in our institution (Gillies, 2016). Due to the highly targeted capabilities of HIFU, whilst leaving superficial skin and pre-focal tissues unharmed, the ablative technology may have a role in treating local recurrence following previous neoadjuvant radiotherapy. For example, following recurrence, HIFU may be able to facilitate conversion from amputation for local control to limb salvage surgery.

Desmoid tumours are a relatively poorly understood subtype of STS which are benign and do not metastasise. However, this tumour subtype demonstrates characteristics of aggressive fibromatosis and comes with significant morbidity and mortality due to their locally invasive nature and, in the familial form, typical bowel involvement. Treatment options are limited and poorly evaluated; mortality is 34% in patients undergoing surgery for intra-abdominal desmoid and post-resection recurrence rates for abdominal wall and intra-abdominal desmoids are 41% and 71% respectively (Sturt, 2006). By virtue of not disrupting the tissue planes, promoting further fibromatosis, HIFU has previously been used on desmoid tumours in small case series outside the UK and have demonstrated encouraging outcomes for both extra- and intra-abdominal desmoid tumours (Shi, 2016), (Ghanouni, 2017).

HIFU is an attractive treatment modality for these indications due to its excellent safety profile, versatility in treating a range of tumour locations (Shim, 2016), its capability to treat multiple smaller tumours in a single session and, furthermore, being repeatable due to the lack of ionising radiation. Oxford has over two-decades of world-class expertise in clinical HIFU with published experiences in translational research of many benign and malignant solid tumour subtypes (Iling, 2005), (Lyon, 2019), (Gilies, 2016), (Leslie, 2012), (Lyon, 2018), (Wu, 2004), (Kennedy, 2004). As the Chinese JC200 device used in Oxford uses diagnostic ultrasound through a water bath to target tumours, rather than an integrated MRI tunnel, treatment of tumours at a variety of anatomical locations becomes both more practical and financially economical.

The clinical HIFU service is complimented by an extensive pre-clinical therapeutic ultrasound research facility at the Institute of Biomedical Engineering, University of Oxford. This laboratory has provided expertise in treatment planning for a previous HIFU clinical trial using patient specific models which employ CT data (Gray, 2019). The multidisciplinary team of co-investigators and other researchers in Oxford have world-class expertise in academic and musculoskeletal radiology, sarcoma surgery, sarcoma radiotherapy and oncology, clinical histopathology and immunology.

Thus, in Oxford there is a unique opportunity to explore the utility of preoperative HIFU in the ablation of infield recurrent STS, smaller STS and desmoid tumours as a pilot study. The primary outcome measure of the study will be safety and feasibility. Radiological response will be explored as a secondary endpoints of efficacy using cross sectional (MRI) and functional imaging (18F-FDG PET), incorporating both size, perfusion and metabolic activity. In addition, novel MRI sequences (DWI including whole body MRI, CEST) may also be explored with the academic radiology department, which pose minimal addition risk to the patient (Chetan, 2019), (Schmidt, 2009).

Crucially, post-resection histology will permit histopathological correlation, mitigating against the possibility of falsely reassuring radiological evaluations (false positive complete ablations). Tertiary endpoints will explore immune response, which HIFU has been demonstrated to mediate (Wu 2004), (Wu, 2016), both through circulating blood markers and immunohistochemistry. This is of importance, as whilst this study may demonstrate safe and effective ablation of targeted STS tumours, there may be micro-metastases or known metastases elsewhere which may limit the overall survival. Thus, thorough understanding of the immune mechanisms at play during HIFU ablation may inform future complimentary systemic treatments. Whilst one other centre has recently published early HIFU experience in STS [6], we believe our proposed study will be the first to elucidate immune mechanisms in HIFU-ablation of STS, and the first trial of HIFU for STS in Europe.

Pain scores and quality of life metrics will also be captured both pre- and post-HIFU and this qualitative data can be used to demonstrate that the HIFU procedure was acceptable to the patient.

ELIGIBILITY:
Inclusion Criteria:

--------

The participant is eligible for the study if they are:

Willing and able to give informed consent for participation in the study.

Aged 18 years or above.

Diagnosed with histologically-confirmed and HIFU-targetable soft tissue sarcoma of several subtypes, including but not necessarily limited to:

* Malignant fibrous histiocytoma
* Undifferentiated (pleomorphic) sarcoma
* Fibrosarcoma and fibromyxoid sarcoma (fibroblastic sarcomas)
* Leiomyosarcoma
* Liposarcoma
* Malignant peripheral nerve sheath tumour
* Retroperitoneal sarcoma
* Rhabdomyosarcoma
* Synovial sarcoma
* Sacral chordoma (following amendment)
* Desmoid tumours (intra- or extra-abdominal, following amendment)

Have at least one of the following:

* Untreated or recurrent primary resectable STS tumour 1-5cm diameter, targetable by HIFU
* Infield recurrent primary resectable STS tumour of >1cm diameter, targetable by HIFU
* Primary or metastatic STS unsuitable for resection or further chemo- or radiotherapy, targetable by HIFU
* Small (1-8cm) symptomatic intra- or extra-abdominal desmoid tumour, targetable by HIFU, which is not indicated for surgery (or patient has declined surgery)

Have life expectancy of over 12 months and a World Health Organisation (WHO) performance status of less than or equal to 1.

Be able to attend Churchill Hospital and Nuffield Orthopaedic Center, Oxford, potentially for multiple visits, and thus be based in the UK.

Willing to allow his or her GP and Consultant to be notified of participation in the study.

Able and willing to give written informed consent, indicating that they are aware of the investigational nature of this study and potential risks, and able to comply with the protocol for the duration of the study, including scheduled follow-up visits and examinations.

Exclusion Criteria:

--------

The participant may not enter the study if ANY of the following apply:

Diagnosed with histologically confirmed Osteosarcoma or Chordoma

Diagnosed with histologically confirmed soft tissue sarcoma of the following subtypes:

* GIST
* Chondrosarcoma
* Kaposi's sarcoma
* Ewings sarcoma
* Giant cell tumour
* Angiosarcoma

Active medical or psychological illness that would render the patient unsuitable for the interventions required for the study (exclusion at the discretion of the investigator).

Pregnancy.

Ulceration / skin breakdown / erythema overlying the target tumour site due to tumour invasion (exclusion at the discretion of the investigator).

Significant radiation skin damage overlying the target tumour site (exclusion at the discretion of the investigator).

Impractical anatomical locations for HIFU targeting (using JC200 treatment device) (exclusion at the discretion of the investigator):

* Retroperitoneum
* Skull
* Neck
* Axilla
* Foot

Unfavourable imaging features on previously acquired cross-sectional imaging, including:

* Tumour within 1cm of the skin surface
* Interposition (or close proximity) of a gas-containing structure between tumour and skin such as fixed (retroperitoneal) bowel or lung
* Interposition of a continuous ossified bone between tumour and skin, such as coverage by pelvis or scapula
* Tumour margin close (<1.5cm) or encasing major neurovascular bundles (such as the sciatic nerve)
* Tumour margin close (<1.5 cm) to critical visceral structures (e.g. bladder or bowel)

Recent radiotherapy (under 6 months) to the target tumour site.

Recent surgery (under 6 weeks) to the target tumour site.

Have any known allergic reactions to intravenous imaging agents to be used in this study (exclusion at the discretion of the investigator).

Have contraindication(s) or intolerance to MRI (exclusion at the discretion of the investigator).

Current involvement in phase 1 studies.

Soft tissue sarcoma participants: Use of chemotherapy or of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the intervention.

Desmoid participants: hormonal medication including the contraceptive pill or tamoxifen, or being treated with imatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse events and serious adverse events deemed due to HIFU | Adverse events endpoint assessed for up to 30 days post-HIFU (or up to point of surgery if sooner)
  Adverse events and serious adverse events deemed due to HIFU recorded using Clavien-Dindo grading
Safety: Number of resectable STS participants converted to unresectable by HIFU | Adverse events endpoint assessed for up to 30 days post-HIFU (or up to point of surgery if sooner)
  Number of resectable STS participants converted to unresectable by HIFU
Safety: Number of limb salvageable STS participants converted to amputation by HIFU | Adverse events endpoint assessed for up to 30 days post-HIFU (or up to point of surgery if sooner)
  Number of limb salvageable STS participants converted to amputation by HIFU
Safety: Number of patients with intra-abdominal desmoid tumour requiring surgery due to complication | Adverse events endpoint assessed for up to 30 days post-HIFU (or up to point of surgery if sooner)
  Number of patients with intra-abdominal desmoid tumour requiring surgery due to complication

SECONDARY OUTCOMES:
Efficacy: Number of resectable STS participants with near pathological complete response | Pathological response assessed within 2 months of surgery or post-HIFU biopsy
  Near pathological complete response (≥95% necrosis) in ≥25% of resectable STS participants post-HIFU
Efficacy: Number of STS participants with non-perfused Volume Ratio (NPVR) Radiological Response | NPVR endpoints assessed using pre-HIFU MRI vs. post-HIFU MRI at: 2-4 weeks (resectable or unresectable), 3-months (±1 month) (unresectable only) and 1-year (±1 month) (unresectable only)
  Non-perfused volume ratio (NPVR) ≥75% on MRI in ≥25% of all STS participants having MRI post-HIFU
Efficacy: Number of STS participants with RECIST Partial Radiological Response | RECIST endpoints assessed using pre-HIFU MRI vs. post-HIFU MRI at: 2-4 weeks (resectable or unresectable), 3-months (±1 month) (unresectable only) and 1-year (±1 month) (unresectable only)
  RECIST partial response in the target tumour alone in ≥25% of unresectable STS participants having MRI post-HIFU
Efficacy: Number of STS participants with PERCIST Partial Metabolic Response | PERCIST endpoints assessed using pre-HIFU MRI vs. post-HIFU PET-CT at: 2-4 weeks (resectable or unresectable), 3-months (±1 month) (unresectable only) and 1-year (±1 month) (unresectable only)
  PERCIST partial metabolic response in the target tumour alone in ≥25% of all STS participants having PET-CT post-HIFU
Efficacy: Number of Desmoid tumour participants with Non-perfused Volume Ratio (NPVR) Radiological Response | NPVR radiological endpoint assessed using pre- and 2-4 weeks post-HIFU MRI
  Non-perfused volume ratio (NPVR) ≥50% on MRI in ≥25% of desmoid participants having MRI post-HIFU
Efficacy: Number of Desmoid tumour participants with RECIST Partial Radiological Response | RECIST radiological endpoint assessed using 1-year post-HIFU MRI
  RECIST partial response in the target tumour alone in ≥25% of desmoid participants having MRI post-HIFU
Efficacy: Number of desmoid tumour and unresectable STS participants with change in Pain Score assessed by Brief Pain Inventory post-HIFU relative to baseline | Pain score and quality of life endpoints assessed at baseline, 2-4 weeks and 3, 6 and 12 months post-HIFU (±1 month)
  Number of desmoid tumour and unresectable STS participants with change in Pain Score assessed by Brief Pain Inventory
Efficacy: Number of desmoid tumour and unresectable STS participants with change in Quality of Life score assessed by EORTC QLQ-C30 | Pain score and quality of life endpoints assessed at baseline, 2-4 weeks and 3, 6 and 12 months post-HIFU (±1 month)
  Number of desmoid tumour and unresectable STS participants with change in Quality of Life score assessed by EORTC QLQ-C30 v3 post-HIFU relative to baseline. In particular Qs 1-28 are on a scale of 1..4 with 1 being best and 4 being worse quality of life.

OTHER OUTCOMES:
Exploratory: Systemic immune effects of HIFU for STS | Tissue samples from baseline (biopsy) and post-surgery stored and analysed with IHC within 6 months. Immune bloods taken at baseline and 2-4 weeks, 3 months, 6 months and 12 months post-HIFU
  To measure the immunological effects of HIFU treatment of STS by immunohistochemistry (IHC) using tumour samples post-HIFU relative to baseline
Exploratory: Local immune effects of HIFU for STS | Tissue samples from baseline (biopsy) and post-surgery stored and analysed with IHC within 6 months. Immune bloods taken at baseline and 2-4 weeks, 3 months, 6 months and 12 months post-HIFU
  To measure the immunological effects of HIFU treatment of STS by immune blood markers using venous blood samples post-HIFU relative to baseline
Exploratory: Number of STS participants with local recurrence within one-year | Within 13 months of HIFU
  One-year local recurrence endpoint assessed using available imaging (CT, MRI, PET-CT)
Exploratory: Number of STS participants with survival for over one-year | Within 12 months of HIFU
  One-year survival endpoint assessed using available clinical information

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Lyon, FRCR, DPhil, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu W, Tang L, Lin F, Jiang L, Shen Z. Significance of HIFU in local unresectable recurrence of soft tissue sarcoma, a single-center, respective, case series in China. Surg Oncol. 2019 Sep;30:117-121. doi: 10.1016/j.suronc.2019.06.004. Epub 2019 Jul 4. PMID 31500773
- [Background] Gillies MJ, Lyon PC, Wu F, Leslie T, Chung DY, Gleeson F, Cranston D, Bojanic S. High-intensity focused ultrasonic ablation of sacral chordoma is feasible: a series of four cases and details of a national clinical trial. Br J Neurosurg. 2017 Aug;31(4):446-451. doi: 10.1080/02688697.2016.1267330. Epub 2016 Dec 12. PMID 27936948
- [Background] Dangoor A, Seddon B, Gerrand C, Grimer R, Whelan J, Judson I. UK guidelines for the management of soft tissue sarcomas. Clin Sarcoma Res. 2016 Nov 15;6:20. doi: 10.1186/s13569-016-0060-4. eCollection 2016. PMID 27891213
- [Background] Tsagozis P, Brosjo O, Skorpil M. Preoperative radiotherapy of soft-tissue sarcomas: surgical and radiologic parameters associated with local control and survival. Clin Sarcoma Res. 2018 Oct 5;8:19. doi: 10.1186/s13569-018-0106-x. eCollection 2018. PMID 30323920
- [Background] Scipione R, Anzidei M, Bazzocchi A, Gagliardo C, Catalano C, Napoli A. HIFU for Bone Metastases and other Musculoskeletal Applications. Semin Intervent Radiol. 2018 Oct;35(4):261-267. doi: 10.1055/s-0038-1673363. Epub 2018 Nov 5. PMID 30402009
- [Background] Illing RO, Kennedy JE, Wu F, ter Haar GR, Protheroe AS, Friend PJ, Gleeson FV, Cranston DW, Phillips RR, Middleton MR. The safety and feasibility of extracorporeal high-intensity focused ultrasound (HIFU) for the treatment of liver and kidney tumours in a Western population. Br J Cancer. 2005 Oct 17;93(8):890-5. doi: 10.1038/sj.bjc.6602803. PMID 16189519
- [Background] Leslie TA, Kennedy JE, Illing RO, Ter Haar GR, Wu F, Phillips RR, Friend PJ, Roberts IS, Cranston DW, Middleton MR. High-intensity focused ultrasound ablation of liver tumours: can radiological assessment predict the histological response? Br J Radiol. 2008 Jul;81(967):564-71. doi: 10.1259/bjr/27118953. PMID 18559903
- [Background] Lyon PC, Rai V, Price N, Shah A, Wu F, Cranston D. Ultrasound-Guided High Intensity Focused Ultrasound Ablation for Symptomatic Uterine Fibroids: Preliminary Clinical Experience. Ultraschall Med. 2020 Oct;41(5):550-556. doi: 10.1055/a-0891-0729. Epub 2019 Jun 25. PMID 31238385
- [Background] Sturt NJ, Clark SK. Current ideas in desmoid tumours. Fam Cancer. 2006;5(3):275-85; discussion 287-8. doi: 10.1007/s10689-005-5675-1. PMID 16998673
- [Background] Shi Y, Huang Y, Zhou M, Ying X, Hu X. High-intensity focused ultrasound treatment for intra-abdominal desmoid tumors: a report of four cases. J Med Ultrason (2001). 2016 Apr;43(2):279-84. doi: 10.1007/s10396-015-0682-9. Epub 2015 Oct 27. PMID 27033872
- [Background] Ghanouni P, Dobrotwir A, Bazzocchi A, Bucknor M, Bitton R, Rosenberg J, Telischak K, Busacca M, Ferrari S, Albisinni U, Walters S, Gold G, Ganjoo K, Napoli A, Pauly KB, Avedian R. Magnetic resonance-guided focused ultrasound treatment of extra-abdominal desmoid tumors: a retrospective multicenter study. Eur Radiol. 2017 Feb;27(2):732-740. doi: 10.1007/s00330-016-4376-5. Epub 2016 May 5. PMID 27147222
- [Background] Shim J, Staruch RM, Koral K, Xie XJ, Chopra R, Laetsch TW. Pediatric Sarcomas Are Targetable by MR-Guided High Intensity Focused Ultrasound (MR-HIFU): Anatomical Distribution and Radiological Characteristics. Pediatr Blood Cancer. 2016 Oct;63(10):1753-60. doi: 10.1002/pbc.26079. Epub 2016 May 19. PMID 27199087
- [Background] Leslie T, Ritchie R, Illing R, Ter Haar G, Phillips R, Middleton M, Bch B, Wu F, Cranston D. High-intensity focused ultrasound treatment of liver tumours: post-treatment MRI correlates well with intra-operative estimates of treatment volume. Br J Radiol. 2012 Oct;85(1018):1363-70. doi: 10.1259/bjr/56737365. Epub 2012 Jun 14. PMID 22700259
- [Background] Lyon PC, Gray MD, Mannaris C, Folkes LK, Stratford M, Campo L, Chung DYF, Scott S, Anderson M, Goldin R, Carlisle R, Wu F, Middleton MR, Gleeson FV, Coussios CC. Safety and feasibility of ultrasound-triggered targeted drug delivery of doxorubicin from thermosensitive liposomes in liver tumours (TARDOX): a single-centre, open-label, phase 1 trial. Lancet Oncol. 2018 Aug;19(8):1027-1039. doi: 10.1016/S1470-2045(18)30332-2. Epub 2018 Jul 11. PMID 30001990
- [Background] Wu F, Wang ZB, Chen WZ, Wang W, Gui Y, Zhang M, Zheng G, Zhou Y, Xu G, Li M, Zhang C, Ye H, Feng R. Extracorporeal high intensity focused ultrasound ablation in the treatment of 1038 patients with solid carcinomas in China: an overview. Ultrason Sonochem. 2004 May;11(3-4):149-54. doi: 10.1016/j.ultsonch.2004.01.011. PMID 15081972
- [Background] Kennedy JE, Wu F, ter Haar GR, Gleeson FV, Phillips RR, Middleton MR, Cranston D. High-intensity focused ultrasound for the treatment of liver tumours. Ultrasonics. 2004 Apr;42(1-9):931-5. doi: 10.1016/j.ultras.2004.01.089. PMID 15047409
- [Background] Gray MD, Lyon PC, Mannaris C, Folkes LK, Stratford M, Campo L, Chung DYF, Scott S, Anderson M, Goldin R, Carlisle R, Wu F, Middleton MR, Gleeson FV, Coussios CC. Focused Ultrasound Hyperthermia for Targeted Drug Release from Thermosensitive Liposomes: Results from a Phase I Trial. Radiology. 2019 Apr;291(1):232-238. doi: 10.1148/radiol.2018181445. Epub 2019 Jan 15. PMID 30644817
- [Background] Chetan MR, Lyon PC, Wu F, Phillips R, Cranston D, Gillies MJ, Bojanic S. Role of diffusion-weighted imaging in monitoring treatment response following high-intensity focused ultrasound ablation of recurrent sacral chordoma. Radiol Case Rep. 2019 Aug 1;14(10):1197-1201. doi: 10.1016/j.radcr.2019.07.004. eCollection 2019 Oct. PMID 31428215
- [Background] Schmidt GP, Reiser MF, Baur-Melnyk A. Whole-body MRI for the staging and follow-up of patients with metastasis. Eur J Radiol. 2009 Jun;70(3):393-400. doi: 10.1016/j.ejrad.2009.03.045. Epub 2009 May 19. PMID 19457631
- [Background] Wu F. Heat-Based Tumor Ablation: Role of the Immune Response. Adv Exp Med Biol. 2016;880:131-53. doi: 10.1007/978-3-319-22536-4_8. PMID 26486336
- [Background] Wu F, Wang ZB, Lu P, Xu ZL, Chen WZ, Zhu H, Jin CB. Activated anti-tumor immunity in cancer patients after high intensity focused ultrasound ablation. Ultrasound Med Biol. 2004 Sep;30(9):1217-22. doi: 10.1016/j.ultrasmedbio.2004.08.003. PMID 15550325
- See also: Sarcoma UK Webpage — https://sarcoma.org.uk/research/focusing-high-intensity-ultrasound-on-sarcoma/